CLINICAL TRIAL: NCT00011193
Title: Dose-response to Exercise in Women Aged 45-75 Years (DREW)
Acronym: DREW
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: PBRC 26043; R01HL066262 (NIH)
Record Dates: First submitted 2001-02-13; First posted 2001-02-13 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Cardiovascular Diseases; Hypertension; Postmenopausal; Overweight or Obese
Keywords: Cardiovascular Diseases; Hypertension; Postmenopausal; Overweight or Obese; Women; Sedentary
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Overweight; Obesity; Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Non-Exercise Control Group: We randomly assigned 102 women in the non-exercise control group and were asked to maintain their level of activity for the 6-month study period.
  Interventions: Behavioral: Exercise
- 4-kcal/kg Energy Expenditure per week: We randomly assigned 155 women to the 4-kcal/kg per week group for 6 months.
  Interventions: Behavioral: Exercise
- 8-kcal/kg Energy Expenditure per week: We randomly assigned 104 women to the 8-kcal/kg per week group for 6 months.
  Interventions: Behavioral: Exercise
- 12-kcal/kg Energy Expenditure per week: We randomly assigned 103 women to the 12-kcal/kg per week group for 6 months.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Compared the effect of 50%, 100%, and 150% of the NIH Consensus Development Panel recommended physical activity dose on fitness in women.

SUMMARY:
To investigate the effects of different amounts of exercise on both cardiorespiratory fitness and risk factors for cardiovascular disease in sedentary, overweight, mildly hypertensive, but healthy, postmenopausal women aged 45 to 75 years.

DETAILED DESCRIPTION:
BACKGROUND:

The primary goal of the Dose-Response to Exercise in Women aged 45-75 Years (DREW) was to investigate the effects of different amounts of exercise on both cardiorespiratory fitness and risk factors for cardiovascular disease. Participants were sedentary, overweight or obese, postmenopausal women who had high normal blood pressure or Stage I hypertension, and thus are at moderately high risk for cardiovascular disease. A total of 464 women (about 35% were recruited from minority groups) were randomly assigned to a control group (N = 102) or to 1 of 3 exercise groups (N = 155 for the lowest exercise dose and 104 in the 8-kcal/kg group and 103 in the 12-kcal/kg exercise group). Women assigned to the exercise groups exercised for 6 months at energy expenditures of 4, 8, or 12 kcal ·kg-1 · week-1. These exercise doses represent the consensus public health recommendation for physical activity from recently published guidelines from the U.S. Public Health Service, American Heart Association, and American College of Sports Medicine (8 kcal ·kg-1 · week-1) and at doses 50% below (4 kcal ·kg-1 · week-1) and 50% above (12 kcal ·kg-1 · week-1) the consensus dose. All women exercised at 50% of V02 max. The exercise sessions took place in the exercise laboratory, with individual supervision of each session and strict control of frequency, duration, and intensity. This was provided thorough documentation of the exact amount of exercise completed. Primary outcome measures are VO2 max and resting systolic blood pressure. Other cardiovascular disease risk factors, psychosocial variables, health-related quality of life, body composition, and fat distribution are secondary outcomes. Other secondary analyses included a focus on the extent to which observed dose-response effects are modified by baseline levels of fitness, ethnicity, risk factors, or age. Assessments will take place at baseline and 6 months. The research provided information about (1) patterns of change in outcomes produced by each of several exercise doses, (2) whether performing exercise at less than the current consensus dose has any benefit, (3) whether performing more exercise than the consensus dose has greater (or proportionally greater) health benefits, and (4) the characteristics of sedentary women who are most likely to benefit from various exercise doses.

DESIGN NARRATIVE:

A total of 464 sedentary, postmenopausal women at moderate risk for cardiovascular disease was randomly assigned to receive exercise training at one of three doses (4, 8, or 12 kcal/kg/wk) or no exercise for six months duration. The specific aims were be to determine: (a) if women in the exercise groups have increased aerobic power (VO2max) over the six months compared to the no exercise group; (b) if women in the exercise groups have a greater reduction in resting systolic blood pressure than those in the no exercise group; and, (c) if there will be a dose-response gradient across the three exercise groups for changes in aerobic power and systolic blood pressure. Secondary aims include evaluating the effects of exercise dose on fasting blood lipids and lipoproteins, glucose, insulin, anthropometry, self-reported quality of life, and cardiovascular risk as determined by a multiple logistic risk function. Covariates to be controlled included dietary intake, physical activity (outside of the exercise program), smoking, alcohol intake, sleep habits, medication use (including hormone replacement therapy), demographics, menstrual history, personal and family medical history.

ELIGIBILITY:
Postmenopausal women aged 45 to 75 years who are overweight or obese (body mass index of 25 to 40 kg/m2) and have normal or mildly elevated BP.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women aged 45 to 75 years who are overweight
Sampling Method: Non-Probability Sample
Enrollment: 464 (Actual)
Dates: Start 2001-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
VO2max and resting systolic blood pressure | at 6 months

SECONDARY OUTCOMES:
Fasting blood lipids and lipoproteins (total, HDL-, and LDL-cholesterol, triglycerides | at 6 months
High sensitive C-reactive protein | at 6 months
Fasting glucose | at 6 months
Anthropometry (body composition and regional fat distribution) | at 6 months
Blood pressure response to exercise | at 6 months
Heart rate variability | at 6 months
Health-related quality of life and other psychosocial variables | at 6 months
Cardiovascular disease risk determined by a multiple logistic risk function | at 6 months
Tertiary Outcomes | at 6 months
  Other variables of interest include dietary habits, physical activity history, smoking, alcohol intake, sleep habits, medication use (including HRT), demographic characteristics, unstructured physical activity, menstrual history, and personal and family medical history.

CONTACTS AND LOCATIONS:
Overall Officials: Steven N. Blair, PED, Principal Investigator — University of South Carolina; Timothy S. Church, MD, PhD, MPH, Principal Investigator — Pennnington Biomedical Research Center; Conrad P. Earnest, PhD, Study Director — University of Bath; James S. Skinner, hD, Study Director — Indiana University
Locations (2):
- United States (2):
  - Oak Cliff-South Dallas, Dallas, Texas
  - The Cooper Institute, Dallas, Texas

REFERENCES:
- [Background] Morss GM, Jordan AN, Skinner JS, Dunn AL, Church TS, Earnest CP, Kampert JB, Jurca R, Blair SN. Dose Response to Exercise in Women aged 45-75 yr (DREW): design and rationale. Med Sci Sports Exerc. 2004 Feb;36(2):336-44. doi: 10.1249/01.MSS.0000113738.06267.E5. PMID 14767260
- [Background] Jurca R, Church TS, Morss GM, Jordan AN, Earnest CP. Eight weeks of moderate-intensity exercise training increases heart rate variability in sedentary postmenopausal women. Am Heart J. 2004 May;147(5):e21. doi: 10.1016/j.ahj.2003.10.024. PMID 15131556
- [Background] Jordan AN, Jurca GM, Locke CT, Church TS, Blair SN. Pedometer indices for weekly physical activity recommendations in postmenopausal women. Med Sci Sports Exerc. 2005 Sep;37(9):1627-32. doi: 10.1249/01.mss.0000177455.58960.aa. PMID 16177618
- [Derived] Kline CE, Sui X, Hall MH, Youngstedt SD, Blair SN, Earnest CP, Church TS. Dose-response effects of exercise training on the subjective sleep quality of postmenopausal women: exploratory analyses of a randomised controlled trial. BMJ Open. 2012 Jul 12;2(4):e001044. doi: 10.1136/bmjopen-2012-001044. Print 2012. PMID 22798253
- [Derived] Johannsen NM, Swift DL, Johnson WD, Dixit VD, Earnest CP, Blair SN, Church TS. Effect of different doses of aerobic exercise on total white blood cell (WBC) and WBC subfraction number in postmenopausal women: results from DREW. PLoS One. 2012;7(2):e31319. doi: 10.1371/journal.pone.0031319. Epub 2012 Feb 17. PMID 22363616
- [Derived] Stewart LK, Earnest CP, Blair SN, Church TS. Effects of different doses of physical activity on C-reactive protein among women. Med Sci Sports Exerc. 2010 Apr;42(4):701-7. doi: 10.1249/MSS.0b013e3181c03a2b. PMID 19952829
- [Derived] Church TS, Martin CK, Thompson AM, Earnest CP, Mikus CR, Blair SN. Changes in weight, waist circumference and compensatory responses with different doses of exercise among sedentary, overweight postmenopausal women. PLoS One. 2009;4(2):e4515. doi: 10.1371/journal.pone.0004515. Epub 2009 Feb 18. PMID 19223984
- [Derived] Martin CK, Church TS, Thompson AM, Earnest CP, Blair SN. Exercise dose and quality of life: a randomized controlled trial. Arch Intern Med. 2009 Feb 9;169(3):269-78. doi: 10.1001/archinternmed.2008.545. PMID 19204218
- [Derived] Earnest CP, Lavie CJ, Blair SN, Church TS. Heart rate variability characteristics in sedentary postmenopausal women following six months of exercise training: the DREW study. PLoS One. 2008 Jun 4;3(6):e2288. doi: 10.1371/journal.pone.0002288. PMID 18523583
- [Derived] Church TS, Earnest CP, Skinner JS, Blair SN. Effects of different doses of physical activity on cardiorespiratory fitness among sedentary, overweight or obese postmenopausal women with elevated blood pressure: a randomized controlled trial. JAMA. 2007 May 16;297(19):2081-91. doi: 10.1001/jama.297.19.2081. PMID 17507344